CLINICAL TRIAL: NCT05206071
Title: Clinical Study of SL19+22 CAR-T Cells for Relapsed or Refractory Non-Hodgkin Lymphoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hebei Senlang Biotechnology Inc., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SL19+22 for NHL
Record Dates: First submitted 2022-01-11; First posted 2022-01-25 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Non-hodgkin's Lymphoma
Keywords: NHL，19+22
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SL 19+22 CAR-T (Experimental)
  Interventions: Biological: CD19+22 CAR-T cells

INTERVENTIONS:
Biological: CD19+22 CAR-T cells — Biological: CD19+22 CAR-T; Drug: Cyclophosphamide,Fludarabine;
  Other Names: CD19+22 CAR-T

SUMMARY:
To evaluate the safety and efficacy of SL19+22 in patients with relapsed or refractory non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
SL19+22 injection is a CAR-T product independently developed by Senlang that targets both CD19 and CD22. Based on the traditional CAR T treatment regimen, the CAR structure was designed, and the activation mode of T cells was changed by using cytokine combination amplification and improved transfection technology.

The Main research objectives:

To evaluate the safety and efficacy of SL19+22 in patients with recurrent or refractory non-Hodgkin's lymphoma

The Secondary research objectives:

To investigate the cytokinetic characteristics of SL19+22 in patients with recurrent or refractory non-Hodgkin's lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent form and be able to comply with the visit, treatment regimen, laboratory examination and other requirements of the study as stipulated in the trial flow chart;
2. The diagnosis of patients with relapsed or refractory non-hodgkin lymphoma;
3. The definition of recurrent or refractory non-Hodgkin lymphoma: Patients with DLBCL, pmbcl and TFL diagnosed by histopathology are resistant to standard treatment; Or PD after at least second-line standard treatment; Or the last treatment effect was SD and the duration was no longer than 6 months; Or CD20 positive patients were ineffective or relapsed after anti-CD20 monoclonal antibody treatment; Or PD after autologous hematopoietic stem cell transplantation or recurrence confirmed by biopsy within 12 months; Or patients undergoing salvage treatment after autologous hematopoietic stem cell transplantation had no remission or recurrence after end-line treatment;
4. There should be at least one measurable tumor foci according to the RECIST version 1.1;
5. ECOG Scores: 0~2;
6. The expression of CD19 and/or CD22 on the tumor cells are reported as positive by either immunohistochemistry or flow cytometry;
7. Estimated survival time is longer than 3 months;
8. Main organ functions shall meet the following requirements: serum creatinine ≤1.5 times the upper limit of normal value (ULN); ALT ULN 2.5 or less; AST ULN 2.5 or less; Total bilirubin ≤ 1.5ULN; Left ventricular ejection fraction (LVEF) ≥45%; Hemoglobin ≥90g/L; Platelet count ≥50×109/L; absolute Neutrophil count (ANC) ≥1.0×109/L; Blood oxygen saturation >92%；
9. Peripheral blood mononuclear immune cells must be collected at least 2 weeks after the last radiotherapy or systemic treatment.

Exclusion Criteria:

1. Serious cardiac insufficiency；
2. Has a history of severe pulmonary function damaging;
3. Coexisting with severe or persistent infection that cannot be effectively controlled;
4. Patients with a history of other malignancies, except those with non-melanoma skin cancer or carcinoma in situ (eg, cervical cancer, bladder cancer, breast cancer) who have received curative treatment at least 2 years prior to screening without disease recurrence;
5. Presence of metabolic diseases (except diabetes and Dyslipidemia);
6. Presence of severe autoimmune diseases or immunodeficiency disease;
7. Patients with active hepatitis B or hepatitis C virus infection;
8. Patients with HIV infection or syphilis infection;
9. Has a history of serious allergies on Biological products (including antibiotics);
10. Participated in any other clinical drug trial for the last three months(except clinicaltrials of CART );
11. Being pregnant, lactating, or planing on pregnancy in the next 12 months.
12. Any situations that the researchers believe will increase the risks for the subject or affect the results of the study(have a history of serious mental illness, drug abuse and addiction).

Ages: 3 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety: Incidence and severity of adverse events | First month post CAR-T cells infusion
  To evaluate the possible adverse events could occurred within first month post infusion.
Efficacy: Overall Remission Rate (ORR) | 3 months post CAR-T cells infusion
  Overall Remission Rate (ORR) including partial remission and complete remission rate after infusion of SL19+22

SECONDARY OUTCOMES:
Efficacy:duration of response (DOR) | 24 months post CAR-T cells infusion
  duration of response (DOR)
Efficacy: progression-free survival (PFS) | 24 months post CAR-T cells infusion
  progression-free survival (PFS) time
CAR-T proliferation | 3 months post CAR-T cells infusion
  the copy number of CD19 and CD22 CAR- T cells in the genomes of PBMC by qPCR
Cytokine release | First month post CAR-T cells infusion
  Cytokine( IL-6,IL-10,IFN-γ,TNF-α ) concentration (pg/mL) by flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Peihua Lu, PhD&M, Principal Investigator — Hebei Yanda Ludaopei Hospital
Locations (1):
- Hebei Yanda Ludaopei Hospital, Langfang, Hebei, China